CLINICAL TRIAL: NCT00660413
Title: Comparison of Acceleromyography and Mechanomyography for Establishing Potency of Neuromuscular Blocking Agents, A Randomized Controlled Study
Brief Title: Comparison of Acceleromyography (AMG) and Mechanomyography (MMG) for Establishing Potency of Neuromuscular Blocking Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: AMG-MMG D-R
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Neuromuscular Blockade
Keywords: Acceleromyography; Mechanomyography; Neuromuscular block; Neuromuscular monitoring; Dose-response; Potency; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG (Experimental): Acceleromygraphy monitoring
  Interventions: Device: TOF-Watch SX (Acceleromyography)
- MMG (Active Comparator): Mechanomyography monitoring
  Interventions: Device: TOF-Watch SX (Acceleromyography)

INTERVENTIONS:
Device: TOF-Watch SX (Acceleromyography) — Randomization of AMG to dominant or non-dominant arm. MMG at contralateral arm.

SUMMARY:
The purpose of this study was to compare two methods for neuromuscular monitoring, acceleromyography and mechanomyography for establishing the dose-response relationship and the potency of a neuromuscular blocking agent using rocuronium as an example. We hypothesized that there would be no significant difference between potencies estimated using acceleromyography and mechanomyography.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Ideal weight +/-20%
* Both arms available for neuromuscular monitoring
* Surgery in supine position
* Participated surgery time more than 30 min

Exclusion Criteria:

* Pregnant and breast-feeding women
* Patients with known illness or use of medications known to influence the neuromuscular transmission
* Known significant renal or hepatic dysfunction
* Allergy to medications used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Comparison of ED50 with the two methods

SECONDARY OUTCOMES:
Comparison of ED95 with the two methods

CONTACTS AND LOCATIONS:
Overall Officials: Casper Claudius, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark